CLINICAL TRIAL: NCT00028327
Title: Randomized Study to Evaluate Immediate Potent Antiretroviral Therapy for HIV-Infected Subjects With CD4 Cell Counts Less Than 350 Cells/mm3 Admitted to Intensive Care Areas With an AIDS-Defining Illness, Pneumonia, or Sepsis
Brief Title: Potent Antiviral Therapy for Critically Ill HIV Infected Patients Admitted to Intensive Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5141; AACTG A5141; A5161s; A5162s
Record Dates: First submitted 2001-12-20; First posted 2001-12-21 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2004-07

CONDITIONS: HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Zidovudine; HIV Protease Inhibitors; CD4 Lymphocyte Count; Lamivudine; Pneumonia; Nelfinavir; Reverse Transcriptase Inhibitors; Antiretroviral Therapy, Highly Active; Efavirenz; Intensive Care Units; Sepsis
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Pneumonia; Sepsis | interventions — lamivudine, zidovudine drug combination; Nelfinavir; efavirenz; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Nelfinavir mesylate
Drug: Efavirenz
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
Many HIV infected patients admitted to the intensive care area (ICA) have never taken anti-HIV drugs. The purpose of this study is to learn whether starting anti-HIV drugs while patients are in an ICA will help them to survive and get better faster. This study will also evaluate patients who, though not in an ICA, have been admitted to the hospital for serious illnesses or infections.

DETAILED DESCRIPTION:
There has been considerable debate over the management of HIV infected individuals admitted to the ICA. Mortality in HIV infected patients in the ICA correlates with the level of immune suppression. The majority of HIV infected individuals entering the ICA are antiretroviral naive. Despite the high mortality rates and the opportunity to intervene with antiretroviral therapy, physicians do not routinely administer highly active antiretroviral therapy (HAART) in the ICA. Early initiation of HAART, which improves immune function, could potentially reduce mortality. Numerous studies have shown that there is a dramatic drop in the HIV-1 RNA levels accompanied by an increase in the CD4 cell count within the first 2 to 4 weeks of therapy. Sufficient data now exist that antiretrovirals could be administered in the ICA with careful monitoring and attention to drug interactions. This study will evaluate the effect of HAART in patients admitted to the hospital with an AIDS-defining illness, pneumonia, or sepsis.

Upon entry into the study, patients are stratified according to a severity of illness score (SAPS I) and CD4 cell count. Patients then are assigned to 1 of 2 study arms: Arm A: HAART (lamivudine [3TC] and zidovudine [ZDV], or 3TC/ZDV, and nelfinavir [NFV] and efavirenz [EFV]); or an alternative HAART for 4 weeks. Arm B: No antiretroviral regimen. Evaluations of the following are performed: drug toxicity, immune status, viral load, arterial blood gas, ventilator parameters, and evolution of the presenting illness. Pharmacokinetic trough concentration analyses are performed on all patients in Arm A during 3 time points of their illness. Patients are followed for 24 weeks after entry. Patients in Arm A may elect to participate in two substudies. The first substudy will measure efavirenz and nelfinavir drug levels in the blood to determine how critical illness affects pharmacokinetics. The second substudy will evaluate the benefit of HAART in HIV infected patients being treated for pneumocystis carinii pneumonia.

ELIGIBILITY:
Inclusion Criteria

* HIV-1 infection
* CD4 cell count less than 350 cells/mm3 within 120 hours prior to study entry
* Admission to an ICA (or to any part of the hospital with an arterial blood gas PaO2/FiO2 ratio of < 200 or SAPS I score > 13) within 120 hours prior to study entry
* Admitted to the hospital for sepsis, pneumonia, or other AIDS-defining disease
* Acceptable methods of contraception

Exclusion Criteria

* Known resistance or intolerance to antiretroviral drugs that precludes use of an effective HAART regimen of FDA approved drugs, excluding abacavir or full-dose ritonavir
* More than 7 days of HAART (a regimen of at least 3 drugs that includes a protease inhibitor, a nonnucleoside reverse transcriptase inhibitor, or three nucleoside analogues) within 4 weeks prior to study entry
* Investigational drug within 14 days prior to study entry
* Pregnant or breast-feeding
* Allergy or sensitivity to any of the study drugs that cannot be substituted with another drug
* CNS mass lesion or bacterial meningitis
* Certain medications
* Uncertain availability for 6 month course of study
* Require regular stomach suctioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Primary Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, Study Chair; Denis Jones, Study Chair
Locations (9):
- United States (9):
  - Univ of Southern California, Los Angeles, California
  - Univ of California, San Diego, San Diego, California
  - Univ of California San Francisco, San Francisco, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Washington Univ School of Medicine, St Louis, Missouri
  - Beth Israel Med Ctr, New York, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Washington, Seattle, Washington